CLINICAL TRIAL: NCT06423404
Title: Video-Guided Active Breaks With Curricular Content on Mental Health and Classroom Climate in Chilean Schoolchildren Aged 6 to 10: Study Protocol for a Multicentre Randomized Controlled Trial
Brief Title: Active Breaks on Mental Health and Classroom Climate in Chilean Schoolchildren Aged 6 to 10
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Concepcion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Universidad de Concepción
Record Dates: First submitted 2024-04-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Mental Health; School-age Children; School Health
Keywords: active break; mental health; school climate; schoolchildren; physical fitness; multicentre randomized controlled trial
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The project involves public primary schools with similar indices of school vulnerability (SVI) and medium to low socioeconomic status in the Biobío province, Chile. This selection was made because students attending these schools spend approximately eight hours per day (from 8:00 AM to 4:00 PM) with two 30-minute breaks and a longer one-hour lunch break. The intervention will focus on 1st to 4th grade classes. Six schools (three treatments and three controls) were recruited, estimating a sample size of 700 students (six schools × eight classes, with each class having 30 to 40 students).
Who Masked: Investigator, Outcomes Assessor
Masking Description: After schools agreed to participate, they were randomly assigned using a sequence generated by the IBM SPSS statistical package, with concealed allocation to one of two groups: 1) the Experimental Group (n=3), receiving a 12-week program of video-guided active breaks with curricular content in the school classroom; and 2) the Control Group (n=3), receiving the same intervention as the experimental group after the final data collection. A simple stratified randomization sequence by sex was used to achieve balance between males and females in both groups. The randomization sequence will be concealed through sequentially numbered, opaque, sealed envelopes, conduct by a project investigator with no contact with schools and participants. Significant differences in the quality of life, motor skills, and academic performance have been found in studies with similar samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Active Break group (Experimental): The Experimental Group, receiving a 12-week program of video-guided active breaks with curricular content in the school classroom
  Interventions: Behavioral: the Experimental Group, receiving a 12-week program of video-guided active breaks with curricular content in the school classroom
- Control group: waiting list group (Other): The Control Group, receiving the same intervention as the experimental group after the final data collection. During the time of the intervention, the waiting list group will receive the usual classes.
  Interventions: Behavioral: the Experimental Group, receiving a 12-week program of video-guided active breaks with curricular content in the school classroom

INTERVENTIONS:
Behavioral: the Experimental Group, receiving a 12-week program of video-guided active breaks with curricular content in the school classroom — The "Active Classes + School Climate and Mental Health" program was crafted following a comprehensive review by the research team on active breaks in the child school population. Based on the findings of this review, the optimal type and duration of intervention, frequency and intensity of the most effective exercises, and video-guided modalities with curricular content for active breaks will be established. Subsequently, a collaborative network was formed, involving researchers from education, sports science, social sciences, medicine, primary school teachers within the Chilean public school system, teams of educational leaders, parents, guardians, pedagogy students, and graduate students. The purpose was to create a team that systematically supports the development of various stages of the project from a multi and interdisciplinary perspective
  Other Names: active break program

SUMMARY:
Background: The incidence of mental health issues in children is increasing worldwide. In Chile, a recent surge in reports of deteriorating mental health among school populations and an increase in complaints related to poor school climate have been observed. Physical activity, specifically active breaks in the classroom, has shown positive effects on children's health. However, evidence regarding its impact on mental health and school climate in children is limited.

Objective: This article outlines the design, measurements, intervention program, and potential efficacy of the Active Classes + School Climate and Mental Health project. This project will assess a 12-week program of active breaks through guided videos with curricular content in the school classroom, and its effects on mental health and school climate as its primary contributions. Additionally, it will measure physical activity, physical fitness, motor competence, and academic performance in students aged 6 to 10 years in the Biobío province, Chile, as secondary contributions.

Methodology: It will be performed a multicenter randomized controlled trial involving students in the 1st to 4th grade (6 to 10 years old), encompassing a total of 48 classes across six schools (three intervention and three control) in the Biobío region, Chile. Video-guided active breaks will be implemented through the Active Classes; web platform, featuring curricular content, lasting 5 to 10 minutes and of moderate to vigorous intensity physical activity, twice a day, Monday to Friday, over a span of 12 weeks.

Expected Results/Discussion: To our knowledge, this will be the first study in Chile to evaluate the effects of incorporating video-guided active breaks with curricular content on mental health variables and school climate in schoolchildren. Thus, this study contributes to the scarce evidence on the effects of video-guided active breaks on mental health variables and school climate in schoolchildren worldwide. Additionally, it will provide crucial information about active teaching methodologies that have the potential to positively contribute to the well-being of students, thus addressing the problems of mental health and climate in Chilean schools.

ELIGIBILITY:
Inclusion Criteria:

- a) Regular male or female students in primary education, from first to fourth grade, at a public school in one of the three provinces of the Biobío region, willing to participate and with parental consent.

b) Students spend at least 38 hours per week in classes (6.5 hours daily) and have at least two short breaks (10-15 minutes) per day.

Exclusion Criteria:

* a) Students with a medical diagnosis of spinal pathologies, vertigo, or uncontrolled hypertension.

  b) Students with severe intellectual disabilities prevented them from following the program instructions.

  c) Students participating simultaneously in another project with similar objectives.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
School climate | From enrollment to the end of treatment at five months
  School climate scale (ECLIS). 82 items with a four-level Likert-type response format (ranging from all to none).
Mental health | From enrollment to the end of treatment at five months
  This outcome will be measurement with School Self-Esteem Test (SSET) and Self-report of socioemotional well-being. The raw score sum is transformed into a T score according to age norms, categorizing students as follows: normal self-esteem, ≥ 40 points; low self-esteem, 30-39 points; and very low self-esteem, ≤ 29 points.

SECONDARY OUTCOMES:
Academic performance | From enrollment to the end of treatment at five months
  The academic performance of the students will be measured using Integral Learning Diagnosis. For this study, only the reading test (2nd, 3rd, and 4th grades) and mathematics test (3rd and 4th grades) were used, measured at the beginning and end of the school year. The grading scale is from 1 as a minimum value to 7 as a maximum value.
Physical health | From enrollment to the end of treatment at five months
  This outcome will be measurement using the Alpha Fitness Test battery protocol, which includes measurements of cardiorespiratory, musculoskeletal, and motor condition.

OTHER OUTCOMES:
Sociodemographic | From enrollment to the end of treatment at five months
  The sociodemographic instrument includes information related to characteristics of the students and their parents (i.e. economic level, educational level). In addition, physical activity and sedentary behavior, eating habits, sleeping and screen habits, type of transportation to the educational center.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Concepción, Concepción, Región del Biobío, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reyes-Amigo T, Ibarra-Mora J, Aguilar-Farias N, Gomez-Alvarez N, Carrasco-Beltran H, Zapata-Lamana R, Hurtado-Almonacid J, Paez-Herrera J, Yanez-Sepulveda R, Cortes G, Rolle-Caceres G, Bezerra A. An active break program (ACTIVA-MENTE) at elementary schools in Chile: study protocol for a pilot cluster randomized controlled trial. Front Public Health. 2024 Jan 8;11:1243592. doi: 10.3389/fpubh.2023.1243592. eCollection 2023. PMID 38259740
- [Derived] Robles-Campos A, Reyes-Molina D, Kracht-Suazo K, Cigarroa I, Carcamo-Oyarzun J, Martinez-Lopez N, Perez-Ruiz M, Grao-Cruces A, Mota J, Ruiz-Ariza A, Munoz Hinrichsen F, Garcia-Perez-de-Sevilla G, Celis-Morales C, Zapata-Lamana R. Effects of Video-Guided Active Breaks on Motor Competence of Schoolchildren with Special Education Needs. Children (Basel). 2025 Jun 21;12(7):820. doi: 10.3390/children12070820. PMID 40723013
- [Derived] Zapata-Lamana R, Robles-Campos A, Reyes-Molina D, Rojas-Bravo J, Salcedo Lagos P, Chavez-Castillo Y, Gajardo-Aguayo J, Villalobos JV, Arias AM, Sanhueza-Campos C, Ibarra Mora J, Reyes-Amigo T, Cristi-Montero C, Sanchez-Oliva D, Ruiz-Hermosa A, Sanchez-Lopez M, Poblete-Valderrama F, Celis-Morales C, Martorell M, Carrasco-Marin F, Albornoz-Guerrero J, Parra-Rizo MA, Cigarroa I. Effects of video-guided active breaks with curricular content on mental health and classroom climate in chilean schoolchildren aged 6 to 10: study protocol for a multicentre randomized controlled trial. Front Physiol. 2024 Sep 12;15:1438555. doi: 10.3389/fphys.2024.1438555. eCollection 2024. PMID 39328832